CLINICAL TRIAL: NCT06708767
Title: Randomized Double Blind Phase 1 Safety Study of CZ10 in Healthy Volunteers
Brief Title: Safety Study of CZ10 in Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nextrast, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: CZ10 Ph 1
Record Dates: First submitted 2024-11-26; First posted 2024-11-27 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteer Study
Keywords: Adverse event; Serious adverse event; safety; intravenous contrast agent; CZ10
MeSH Terms: interventions — Contrast Media

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low dose (Experimental): 400 mg/kg CZ10 intravenous administration
  Interventions: Drug: Contrast Media; Drug: Placebo
- Medium dose (Experimental): 800 mg/kg CZ10 intravenous administration
  Interventions: Drug: Contrast Media; Drug: Placebo
- High dose (Experimental): 1200 mg/kg CZ10 intravenous administration
  Interventions: Drug: Contrast Media; Drug: Placebo

INTERVENTIONS:
Drug: Contrast Media — IV contrast media administration
Drug: Placebo — Saline

SUMMARY:
A randomized, double-blind, placebo-controlled, parallel group, dose escalation study in healthy subjects to evaluate the safety, tolerability, pharmacokinetics and initial effectiveness of a novel intravenous CT contrast material (CZ10).

This first-in-human clinical phase 1 trial will test the safety of escalating doses of CZ10 that has shown high safety and efficacy as a intravenous contrast agent in preclinical trials.

The subjects for this study will be healthy adult volunteers, including obese but otherwise healthy subjects up to 450 lbs or the maximum allowable weight of the CT scanner, whichever is lighter. Subjects will be recruited and randomly assigned to cohort and test article.

A total of 24 subjects will be evaluated with 18 subjects randomized to receive active drug and 6 subjects randomized to receive placebo control in a double blind manner. A total of three cohorts of 8 subjects will be enrolled. The first cohort subjects will receive a low dose, then if less than 2 subjects show severe adverse events, the second cohort will receive the expected clinical dose, then if less than 2 subjects show severe adverse events, the last cohort will receive a high dose of the intravenous test article. For each cohort, six subjects will be randomized to receive CZ10 and two to placebo. To increase subject safety, two initial subjects from each cohort will be randomized one to receive CZ10 and the other to receive placebo. If there are no serious adverse events through 3 days post dosing, then the remainder of the cohort will be enrolled.

Subjects will be screened and enrolled up to 30 days prior to the day of test article dosing. Inclusion criteria are adult subjects willing to consent for the trial. Exclusion criteria are persons: (a) who are pregnant (as determined by a urine pregnancy test at the time of consent); (b) who have significant cardiovascular, respiratory, hepatic, gastrointestinal, hematological, neurological, psychiatric or other disease that may interfere with the objectives of the study and/or pose safety concerns; (c) Have evidence of moderate to severe renal insufficiency or renal failure (defined as an estimated glomerular filtration rate <60 ml/minute); (d) who have an allergy to iodinated CT or other medical intravenous contrast material; (e) who are more than 450 pounds which would result in inability to be scanned on CT; or (f) have poor venous access such that an 18g venous cannula cannot be placed into the antecubital or other large superficial arm vein. Exclusion criteria also include women who are breastfeeding and women of childbearing age who are not using double protection birth control.

Safety assessments will include monitoring of adverse events, vital signs (blood pressure, pulse rate, respiratory rate and oral temperature), clinical laboratory findings, 12-lead ECGs, subject reporting of symptoms, and physical examination findings. A physical examination will be performed at screening and on Day 2 and Day 7. A resting 12-lead ECG will be performed at screening, pre-dose and on Day 1 at 4 hours, Day 2, and Day 7. Vitals signs will be assessed at screening, at admission to the clinical research unit the day of dosing, then at 2, 4, and 7 hours after dosing, and on Day 2 and Day 7. Clinical laboratory tests (chemistry and hematology) will be performed at screening, pre-dose, at 7 hours after start of oral dosing, and Day 2 and 7 after dosing. A phone call interview to assess for symptoms will occur on day 15. In particular subjects will be monitored for possible allergic reaction, contrast material extravasation, and possible renal injury. If any adverse events are seen, the subject will be return to the clinical research unit for further assessment and possible treatment.

Tentatively, the doses of CZ10 are expected to be 400, 800, and 1200 mg / kg of CZ10 but final doses will depend on preclinical and manufacturing data. The dose of test article will likely be limited by volume of material that can be bolus injected (maximum feasible dose). The placebo will be given at the same dose volume as the CZ10 drug product.

At the conclusion of the study, the necessary safety data will be available to decide on whether and how to proceed with clinical phase 2 studies on patients with suspected or known vascular disease.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled, parallel group, dose escalation study in healthy subjects to evaluate the safety of intravenous CZ10 medical imaging contrast material.

Development of a new intravenous clinical CT contrast agent would provide diagnostic value for CT, particularly for patients unable to tolerate existing agents. The current study will be the first-in-human test of a novel CZ10 contrast material with excellent signal and safety in preclinical testing.

Supporting Preclinical Safety Data

CZ10 has been the subject of substantial in vivo and safety research. CZ10 undergos renal elimination with low retention in other organs, comparable to those of current CT contrast agents. CZ10 is well tolerated, having been administered to rats at 3000 mg/kg, and repeatedly in rabbits and pigs at 400 - 540 mg/kg. CZ10 showed minimal, transient increase in only one urinary kidney stress marker (neutrophil gelatinase-associated lipocalin, NGAL) after 1500 mg/kg IV injection in rats, but no histopathological evidence of kidney injury was seen. Blood counts and clinical chemistry of rats given CZ10 at 1500 and 3000 mg/kg were unchanged from controls. Blood counts and clinical chemistry measurements from rabbits and swine also showed no adverse effects, although these studies were imaging-focused where safety was not an endpoint. Peritoneal injection of CZ10 at 500 mg/kg in rats showed rapid clearance at CT imaging on day 2 with no observable toxicity. Good laboratory practice testing of CZ10 in rat and dog showed no toxicity referable to CZ10.

INVESTIGATIONAL PLAN

OVERALL STUDY DESIGN

This is a randomized, double-blind, placebo-controlled, parallel group, dose escalation study in healthy subjects to evaluate the safety of intravenous CZ10 CT contrast material.

This first-in-human clinical phase 1 trial will test the safety of escalating doses of CZ10 that has shown high safety and efficacy as an intravenous contrast agent in extensive preclinical testing.

The subjects for this study will be healthy adult volunteers, including obese but otherwise healthy subjects up to 450 lbs. Subjects will be recruited and randomly assigned to cohort and test article.

A total of 24 subjects will be evaluated with 18 subjects randomized to receive active drug and 6 subjects randomized to receive placebo control in a double blind manner. A total of three cohorts of 8 subjects will be enrolled. The first cohort subjects will receive a low dose. A review of safety data from all 8 subjects will be performed. If less than 2 subjects show severe adverse events, then the second cohort will be enrolled. A review of safety data from these 8 subjects will then be reviewed, and if less than 2 subjects show severe adverse events, the last cohort will be enrolled. This last cohort will receive a high dose of the intravenous test article. For each cohort, six subjects will be randomized to receive CZ10 and two to placebo.

The study will be performed at a dedicated Clinical Phase 1 center. A dedicated Clinical Phase 1 center is desirable due to the specialized testing and subject recruitment required and the need for strict adherence to the procedures in the study manual. Good clinical practice will be emphasized and documented for all aspects of this trial.

INVESTIGATIONAL PRODUCT - INJECTABLE CONTRAST

Investigational Product and Placebo Description CZ10 will be administered as an injectable formulation. The aqueous formulation will have been prepared as a sterile bottled transparent fluid. A similar appearing saline placebo will be prepared.

Investigational Product Preparation The bottle of the agent will be opened in the CT suite and loaded manually into the CT injector syringe in the same manner as conventional CT contrast material, with care to remove gas bubbles. The volume of injection is likely to be 2 mL per kg body weight, but may be increased to 5 mL per kg of body weight in the high dose group. In some obese subjects, a dose volume of 2 or 4 mL per kg may not be achievable due to limitations of the contrast power injector. In such cases, the maximum feasible dose will be used (the limit of the power injector, which is 220 mL). This adjustment and maximum dose volume reflects standard practice in clinical radiology.

Investigational Product Storage and Accountability Investigational product will be stored at room temperature in a secure, locked area, under the responsibility of the clinical research unit pharmacy or its designee. The Investigator or Investigational Pharmacy must maintain accurate records of the receipt of all study drug, including date received, lot number, amount received, condition of the package and the disposition. Dispensing records will be maintained including the date and amount of study drug dispensed and the identity of the subject receiving the study drug.

Following dosing, all empty bottles will be retained until reconciliation with the dispensing and shipping records is complete. Empty bottles may then be destroyed per investigative pharmacy policy.

Following final reconciliation (at the end of the study), unused study drug may either destroyed according to site guidelines or returned to Nextrast, Inc.

Investigational Product Packaging and Labeling Labels will be accordance with all applicable regulatory requirements for the labeling of active pharmaceutical ingredients. Labels will contain the drug name, protocol number, date of manufacture, storage conditions and a caution statement that the drug is for clinical investigational use only.

Methods of Assigning Subjects to Dose Groups:

The subject treatment assignment will be based on a computer generated randomization scheme with a ratio of 3:1 (active:placebo) for each of the three drug level cohorts. The study drug blind will be maintained through a randomization schedule held by the Pharmacist randomization personnel in the CRU pharmacy.

SUBJECT POPULATION

Inclusion Criteria

To be eligible for enrollment, a subject must meet the following criteria:

1. Understands the requirements of the study and provides written informed consent prior to undergoing any study-related procedures
2. Subject is between the ages of 18 to 85 years old, inclusive
3. Has good venous access as determined by the Investigator at screening
4. Is able to lie flat with arms above head for 15 mintues and hold breath for 15 seconds
5. Weighs up to 450 lbs

Exclusion Criteria

Subjects will be excluded from the study if they meet any of the following criteria:

1. Is pregnant (as determined by a urine pregnancy test at the time of consent)
2. Has significant cardiovascular, respiratory, hepatic, gastrointestinal, hematological, neurological, psychiatric or other disease that may interfere with the objectives of the study and/or pose safety concerns;
3. Has evidence of moderate to severe renal insufficiency or renal failure (defined as an estimated glomerular filtration rate <60 ml/minute)
4. Has an allergy to iodinated CT or other medical intravenous contrast material
5. Weighs more than 450 pounds which would result in inability to be scanned on CT
6. Is breastfeeding
7. Is a woman of childbearing age who is not using double protection birth control

Replacement of Subjects This study plans to enroll 24 evaluable subjects. For the purpose of this study "evaluable" subjects are those that are successfully injected with the full dose of intravenous test article. Non-evaluable subjects may be replaced following discussion between the Principal Investigator and Nextrast.

SCHEDULE OF PROCEDURES

Study Visits There are 4 planned in-clinic visits and 1 planned follow-up phone call for this study. Additional visits may be needed if follow up for an adverse event is needed or if screening cannot take place in a single visit. Investigators should schedule visits within the protocol-specified timelines unless they receive permission from Nextrast, or unforeseeable events prevent the subject from complying.

All study procedures must be recorded in source documentation (primary occurrence of a record) maintained by the clinical site.

Informed Consent Prior to performing any study-related activities under this protocol, including screening tests and assessments, written informed consent with the IRB-approved ICF must be obtained from the subject in accordance with local practice and regulations.

A copy of the ICF, signed and dated by the subject, must be given to the subject and documented in the subject's source documentation. The original signed consent form will be retained with the study records

Screening Visit (Days -30 to 0):

Once informed consent is obtained, the following assessments will be done to establish a subject's eligibility for the study. Note: in cases where subjects have given consent for general pre-screening at the site, some of these assessments may be done via chart review.

When possible, the assessments should be done in the order listed here to avoid the demands of sample collection and ECG prior to the subject passing basic entry criteria requirements.

* Review of eligibility requirements - inclusion and exclusion criteria
* Collection of demographic information and medical history, including review of prior and ongoing medications (taken in previous 30 days)
* Limited Physical Exam
* Vital signs measurement (blood pressure, pulse rate, respiratory rate and oral temperature)
* In women of child-bearing potential, urine sample for pregnancy test Once eligibility is established, subjects will be scheduled for their Day 1 visit

Day 1 Visit: Dosing and Imaging

Subjects will be instructed to arrive early in the morning to the clincal research unit. The following assessments must be done in the order noted:

1. Pre-dose: May be done up to 2 hours before start of dosing

   * Review eligibility and update of medical history as needed
   * Conduct 12-lead ECG
   * Take vital signs (BP, PR, RR, temperature)
   * Obtain blood and urine samples for clinical laboratory tests
   * Obtain blood and urine samples for PK
   * Place arm venous catheter (at least 20g)
2. IV Dose Administration:

   o Given via venous catheter in arm
3. Post-dosing: Approximately 4 hours post dose

   * Conduct 12-lead ECG
   * Take vital signs (BP, PR, RR, temperature)
   * Obtain blood and urine samples for clinical laboratory tests
   * For subjects in the PK subgroup: obtain blood and urine samples for PK
   * Query subjects for possible AEs Subject may be discharged from the clinic with instructions to return the next day for the Day 2 visit. Subjects should be reminded to make note of any changes in their health that will be reviewed by the investigator at the Day 2 visit.

Day 2 Visit: In-clinic Follow-up or Early Termination

The following assessments are included in this visit and may also be done if a subject withdraws from the study early:

* Limited physical exam
* 12-lead ECG
* Vital signs (BP, PR, RR, temperature)
* Obtain blood and urine samples for clinical laboratory tests
* For subjects in the PK subgroup: obtain blood and urine samples for PK
* Query subjects for possible AEs If the investigator has no further concerns which require medical attention or follow up, the subject may be released from the clinic with a reminder that they will need to return on Day 7.

Day 7 Visit: In-clinic Follow-up or Early Termination

The following assessments are included in this visit and may also be done if a subject withdraws from the study early:

* Limited physical exam
* 12-lead ECG
* Vital signs (BP, PR, RR, temperature)
* Obtain blood and urine samples for clinical laboratory tests
* Query subjects for possible AEs If the investigator has no further concerns which require medical attention or follow up, the subject may be released from the clinic with a reminder that they will receive a phone call from the clinic on Day 15 +/-2 days, to inquire about any changes in their health since this follow-up visit.

Day 15 ± 2: Telephone follow up Every subject who has completed the study through the Day 7 visit, will be called by a member of the site study staff on Day 15 +/-2 days. The purpose of the call is to determine if any new health issues have arisen that may require follow up in the clinic by the Investigator or designee. New health issues reported by the subject should be reviewed with by the Investigator who will determine whether or not they constitute a new adverse event. The caller should also establish whether any AEs ongoing at the time of the Day 7 visit have resolved. If not, the Investigator should be informed, and a determination made whether or not more follow up is needed.

EARLY DISCONTINUATION/WITHDRAWAL PROCEDURES The entire study may be discontinued at the discretion of Nextrast. In these circumstances the Investigator will arrange for a final visit for those subjects not having reached Day 2 or 7 and a follow-up phone call for those subjects having completed the Day 7 visit but not the Day 15 phone call.

Subjects are free to withdraw from study participation at any time, for any reason, and without prejudice.

The participation of an individual subject in the study may be terminated in the following circumstances:

1. Withdrawal of informed consent by the subject
2. Inability to complete dosing with the IV contrast
3. Any occurrence that, in the Investigator's opinion, makes continued participation contrary to the subject's best interests.

   If an investigator removes a subject from the study, or if a subject declines further study participation, an Early Discontinuation Visit, consisting of the assessments required at the Day 2 or 7 visit, will be completed as soon as possible. It will be the responsibility of the Investigator to ensure that all withdrawn subjects receive appropriate follow-up and medical care if needed.

   SAFETY ASSESSMENTS

   Assessment of Safety:

   Safety will be assessed by the recording of adverse events, vital signs, changes in physical exam, 12-lead ECGs and the following clinical laboratory tests:

   Hematology
   * Hemoglobin (Hgb)
   * Hematocrit (Hct)
   * Platelet count
   * Red blood cell count
   * White blood cell count with differential

   Chemistry
   * Blood Urea Nitrogen (BUN)
   * Creatinine
   * Total bilirubin
   * Alkaline Phosphatase
   * Aspartate transaminase (AST)
   * Alanine transaminase (ALT)
   * Gamma-glutamyl transferase (GGT)
   * Lactic dehydrogenase (LDH)
   * Glucose
   * Albumin
   * Total protein
   * Bicarbonate
   * Phosphate
   * Sodium
   * Potassium
   * Chloride
   * Calcium
   * Total cholesterol
   * Urate

   Urinalysis
   * pH
   * Specific gravity
   * Protein
   * Glucose
   * Ketones
   * Bilirubin
   * Blood
   * Nitrites
   * Leukocytes
   * Urobilinogen
   * Microscopic urine analysis

   Adverse Events Adverse event solicitation and recording will begin immediately following dosing with the study product (CZ10 IV contrast) and will include only on-treatment (treatment emergent) events. Any changes to a subject's health that occur between the signing of the informed consent and dosing will be recorded as updates to the subject's medical history.

   Subjects will be instructed to report AEs during the study and staff will query subjects regarding AEs throughout the study. The Investigator (and/or designee) must document all AEs reported from the time of dosing through completion of the Day 15 phone call. Any subject who is withdrawn from the study due to an AE shall be followed until the event has resolved or stabilized or 15 days after last dose and the Investigator will document available follow-up information on the subject's source documentation and CRF

   Definition of an Adverse Event NOTE: The Investigator's Brochure contains safety information for CZ10 obtained from the preclinical studies An adverse event (also referred to as an adverse experience) can be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug and does not imply any judgment about causality. An adverse event can arise with any use of the drug (e.g., off-label use, use in combination with another drug) and with any route of administration, formulation, or dose, including an overdose.

   Adverse Events are NOT:
   * Medical or surgical procedures (e.g., surgery, endoscopy, tooth extraction, transfusion). The condition that leads to the procedure is the AE.
   * Situations where an untoward medical occurrence has not occurred (e.g., hospitalization for elective surgery, social and/or convenience admissions).
   * Worsening of symptoms associated with expected decline in the disease being studied by CT.

   Evaluating and Reporting of Adverse Events All AEs (i.e. a new event or an exacerbation of a pre-existing condition) that occur after dosing with NX9 and up to 14 days post-dosing must be recorded as an AE or SAE (if applicable), on the Adverse Event eCRF and SAE form, as applicable. The Investigator must follow all AEs until the AE resolves, or until the Investigator and/or the Medical Monitor determine the event is chronic or clinically stable. If an AE remains unresolved at the conclusion of the study, the Investigator and Medical

   Monitor will make a clinical assessment to determine whether continued follow-up of the AE is warranted. All subjects who have received at least one exposure to study therapy will be evaluated for safety of study treatment.

   The Investigator should attempt to establish a diagnosis of the event based on signs, symptoms and/or other clinical information. In such cases, the diagnosis should be documented as the AE and not the individual signs/symptoms.

   All AEs must be promptly documented on the Adverse Event eCRF and assessed by the Investigator. Details of the event must include the dates of onset and resolution, severity, relationship to study drug, seriousness, and whether the event caused the subject to withdraw from the study, outcome and timing with regard to administration of the study drug.

   Severity: Severity should be graded and recorded as follows:
   * Mild: Awareness of event but easily tolerated
   * Moderate: Discomfort enough to cause interference with usual activity
   * Severe: Inability to carry out usual activity, incapacitating, requires medical intervention

   Relationship: The relationship of the Adverse Event to the study drug will be determined by the Principal Investigator, and assessed using the following definitions:
   * Related: There is a distinct temporal relationship between the event onset and administration of the study drug. There is a known reaction to agent or chemical group or predicted by known pharmacology. The event cannot be explained by subject's clinical state or other factors.
   * Unrelated: Evidence exists that the AE has an etiology other than the study drug (e.g., pre-existing condition, underlying disease, intercurrent illness, or concomitant medication).

   These criteria, in addition to good clinical judgment, should be used as a guide for determining the causal assessment. If it is felt that the event is not related to study drug therapy, then an alternative explanation should be provided.

   Serious Adverse Events (SAEs) All SAEs as defined below and that occur after the first dose of Z10 and up to 15 days post-dose must be reported to Nextrast as soon as the site becomes aware of them. Any SAEs occurring more than 15 days after last study drug administration and considered at least possibly drug-related must also be reported.

   An SAE is an AE from this study that results in any of the following outcomes:
   * Death
   * Life-threatening situation (subject is at immediate risk of death)
   * Inpatient hospitalization or prolongation of existing hospitalization
   * Persistent or significant disability/incapacity
   * Congenital anomaly/birth defect in the offspring of a subject who received study drug

   NOTE: Important medical events that may not result in death, be immediately life- threatening, or require hospitalization, may be considered an SAE when, based upon appropriate medical judgment, they may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

   A life-threatening AE is defined as any adverse experience that places the subject in the view of the Investigator, at immediate risk of death from the event as it occurred. This does not include an event that might have led to death, if it had occurred with greater severity.

   "Inpatient hospitalization" means the subject has been formally admitted to a hospital for medical reasons, for any length of time. Presentation and care within an emergency department does not necessarily constitute an SAE. Complications that occur during hospitalization are AEs. If a complication prolongs hospitalization, it is an SAE.

   All deaths, regardless of cause, must be reported for subjects on study (within 28 days of last study drug dose). The SAE term should reflect the event that leads to the death with "death" recorded as the outcome

   Clinical Laboratory Abnormalities and Other Abnormal Assessments Laboratory abnormalities are usually not recorded as AEs unless considered to be clinically significant by the site clinician. An abnormal laboratory result will be considered an AE if it induces clinical signs or symptoms, if the abnormality is of a degree that requires active management (e.g. discontinuation of the study drug, dose modification) or when the event is requiring treatment or other therapeutic intervention (e.g. iron supplements, blood transfusion, etc.).

   The Investigator will evaluate the relationship of any significantly abnormal result to protocol treatment and clinical condition, if possible. All clinically significant abnormal laboratory results will be followed until they return to normal or become stabilized.

   Safety assessments of particular concern:

   While safety assessments will be open ended, particular attention will be made to possible allergic reaction, renal injury, and contrast material extravasation. This concern is because these adverse events have been associated with intravenous contrast material. Monitoring for these adverse events will be as follows:

   i) Allergy. Subjects will be monitored during injection of the intravenous agent, at time of procedure, when they leave, and by phone/follow-up visit thereafter.

   ii) Renal injury. Subjects will be monitored by serial serum creatinine and urinalysis including 1 and 7 days after injection of the contrast material, and by phone/follow-up visit thereafter. Any patients reporting hematuria, oliguria, swelling of the legs, or other symptoms that may be related to renal insufficiency will be asked to return to visit with study personnel for further investigation.

   iii) Subcutaneous extravasation of contrast material. Subjects will be monitored during and immediately after injection of the intravenous contrast agent for signs of local extravasation of contrast material. If contrast material extravasation is suspected, then that body part will be massaged, treated with cold compress, and elevated. The body part and the distal arm and fingers will be monitored for pain, numbness, and strength. If there is concern for compartment syndrome, the subject will be transferred to the emergency department to be monitored for elevated compartmental pressures and will be assessed by emergent plastic surgery consultations.

   STATISTICAL METHODS

   STATISTICAL METHODS

   General Considerations All quantitative endpoints will be summarized using descriptive statistics (n, mean, standard deviation, median, 25th quartile, 75th quartile, minimum and maximum values). All qualitative endpoints will be summarized by the number of subjects meeting the endpoint and the percentage of subjects out of the appropriate population. The denominator will be displayed when needed.

   Statistical inference will be performed as appropriate. Only two-sided tests with an α=0.05 will be used.

   Analysis Populations

   The following analysis populations are planned:

   • Safety Population: All subjects who receive an administration of NX9 contrast.

   Subject Disposition and Demographic Data The number of subjects screened and treated will be summarized. The denominator for the calculation of percentages will be from the number of subjects treated.

   The following categories will also be summarized for subject disposition:
   * Completed the study
   * Discontinued from the study early and the reason for discontinuation Subject demographics will be summarized for all subjects in the safety population. Appropriate baseline characteristics will be included in addition to demographic characteristics. No statistical testing will be performed. Additional details will be provided in the Statistical Analysis Plan (SAP).

   Safety Endpoints Safety will be evaluated by assessment of clinical laboratory tests, PE, ECG and vital signs measurements at various time points during the study, and by the documentation of AEs. All safety data collected on or after administration of NX9 contrast will be summarized.

   All data collected during the course of the study will be included in the data listings.

   Adverse Events Adverse events will be summarized by the Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term. All subjects in the safety analysis set will be included in the summaries. Events will be summarized on the basis of the date of onset for the event. A treatment-emergent adverse event (TEAE) will be defined as any adverse event that begins on or after the date of administration of NX9 contrast.

   An overall summary of TEAEs will be provided. Summaries (number and percentage of subjects) of TEAEs (by System Organ Class and Preferred Term) will be provided:
   * TEAEs
   * Treatment-related TEAEs
   * TEAEs leading to study drug discontinuation
   * Serious TEAEs
   * Treatment-related Serious TEAEs

   No statistical testing will be performed. All AEs collected during the study will be presented in the data listings. Additionally, a listing will be provided for any AEs leading to death.

   Clinical Laboratory Data Summaries of clinical laboratory results and change from baseline will be performed using descriptive statistics by visit. All subjects in the safety population will be included in these summaries. No statistical testing will be performed.

   Other Safety Evaluations Individual data for physical examination findings, prior and concomitant medications and medical history will be provided. Twelve-lead ECGs and vital signs measurements will be listed by subject and summarized by incidence of events/abnormalities or descriptive statistics as appropriate. No statistical testing will be performed.

   CRITERIA FOR STUDY TERMINATION The Investigator has the right to terminate the study in the interest of subject safety and welfare in consultation with Nextrast, Inc. Nextrast, Inc. reserves the right to terminate or amend the study at any time for administrative reasons or if continuation of the protocol would present a potential safety risk to the subjects.

   PROHIBITIONS AND RESTRICTIONS

   Subjects must be willing to adhere to the following prohibitions and restrictions during the entire course of the study:
   * No consumption of alcohol or food containing alcohol,
   * No administration of any prescription drugs,

   SUBJECT WITHDRAWAL CRITERIA Subjects will be informed that they have the right to withdraw from the study at any time for any reason without prejudice to their medical care. The Investigator also has the right to withdraw subjects from the study if it is in the best interest of the subject, or if the subject experiences an adverse event that warrants premature withdrawal.

   Subjects may be withdrawn from the study if they:
   * Have entered the study in violation of the protocol
   * Use or require the use of prohibited concomitant medication(s)
   * Are non-compliant with study procedures
   * Experience an AE that warrants premature withdrawal

   All treated subjects, should be followed according to the Schedule of Procedures above. All subjects, even those who have discontinued prematurely, should have all evaluations for the End-of-Study visit performed, if possible. All procedures and the subjects' final disposition should be documented in the case report form (CRF). For all subjects who withdraw prematurely, the Investigator will indicate one of the following reasons for withdrawal on the Clinical Research Form:
   * Death
   * Lost to Follow-up
   * Adverse Event
   * Non-Compliance with Study Drug
   * Physician Decision
   * Pregnancy
   * Protocol Violation
   * Study termination by Sponsor
   * Withdrawal of Consent

   Any subject who discontinuations from the study due to an AE will be closely monitored until the resolution or stabilization of the AE or until 30 days after last dose, whichever occurs first. The Investigator should document the reason for discontinuation in the source documentation and CRF.

   In the event that a subject withdraws consent for study participation, early withdrawal should be documented by the Investigator (or designee) in the appropriate CRF pages and source documents when confirmed.

   Early Withdrawal Visit:

   As outlined above, in the event that a subject discontinues study participation at any time prior to the final End-of-Study phone call, if possible, the subject should complete all follow-up assessments, as described for Day 2. The reason for discontinuation must be fully documented in the subject's source documentation and in the clinical research form.

   BLINDING This study is a double-blind study, meaning that the subjects and investigators will not know whether the subjects are being dosed with active or placebo study product. This double blind approach helps ensure objectivity in assessments. The clinical site pharmacist or designee will serve as the randomization holder and will dispense both active drug and placebo on the day of administration according to the randomization schedule.

   Randomization data are kept strictly confidential and are accessible only by authorized personnel and emergency codes will be available to the pharmacy which reveal the treatment group assignment for a specific study subject that may be opened during the study only if the subject's well-being requires knowledge of the subject's treatment assignment. If the investigator decides that unblinding is warranted, the investigator should make every effort to contact the Nextrast (Medical Monitor, or Representative) prior to unblinding a study subject's treatment assignment. When a study subject's treatment assignment is unblinded Nextrast, Inc. should be notified immediately.

   The investigation's drug blind shall not be broken by the PI unless information concerning the investigational drug is necessary for the medical treatment of the subject. All study assessment and causality should be performed if possible before unblinding. In the event of a medical emergency, if possible, the MM or designee should be contacted before the investigational drug blind is broken to discuss the need for unblinding. The sponsor must be notified as soon as possible if the investigation drug blind is broken.

   The investigational drug blind shall not be broken by the PI unless information concerning the investigational drug is necessary for the medical treatment of the subject. All study assessment and causality should be performed if possible before unblinding. In the event of a medical emergency, if possible, the Medical Monitor or designee should be contacted before the investigational drug blind is broken to discuss the need for unblinding. The sponsor must be notified as soon as possible if the investigation drug blind is broken. The subject blind can be broken only if the Principal Investigator deems it necessary for the safety of the subject and preferably after consulting with the Medical Monitor at Nextrast, Inc. The blind may be broken for an individual subject who meets dose escalation stopping criteria during

ELIGIBILITY:
Inclusion Criteria:

* Understands the requirements of the study and provides written informed consent prior to undergoing any study-related procedures
* Subject is between the ages of 18 to 85 years old, inclusive
* Has good venous access as determined by the Investigator at screening
* Weighs up to 450 lbs

Exclusion Criteria:

* Is pregnant (as determined by a urine pregnancy test at the time of consent)
* Has significant cardiovascular, respiratory, hepatic, gastrointestinal, hematological, neurological, psychiatric or other disease that may interfere with the objectives of the study and/or pose safety concerns;
* Has evidence of moderate to severe renal insufficiency or renal failure (defined as an estimated glomerular filtration rate <60 ml/minute)
* Has an allergy to iodinated or other medical intravenous contrast material
* Weighs more than 450 pounds
* Is breastfeeding
* Is a woman of childbearing age who is not using double protection birth control

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2050-01 (Estimated); Primary Completion 2052-01 (Estimated); Study Completion 2054-01 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events | Within 2 weeks after dosing with intravenous contrast material
  Number of adverse event cases reported
Abnormality cases in lab test results | Within 1 week after dosing with intravenous contrast agent
  Number of clinically significant abnormalities found in lab test results.
Abnormality cases physical exam results | Within 1 week after administration of intravenous contrast agent
  Number of clinically significant abnormalities found in physical exam results
Abnormality cases in vital signs | within 1 week after administration of IV contrast agent
  Number of clinically significant abnormalities found in vital signs
Abnormality cases in 12-lead ECG | Within 1 week after dosing with intravenous contrast agent
  Number of clinically significant abnormalities found in 12-lead ECG